CLINICAL TRIAL: NCT00958919
Title: The Role of Endorphins in the Perception of Dyspnea With Resistive Loading in Patients With COPD
Brief Title: Role of Endorphins in Perception of Dyspnea With Resistive Loading in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21721
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Results first posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: breathlessness intensity; breathlessness unpleasantness; endorphins; resistive breathing loads
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Naloxone; Saline Solution; Fluoridation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- naloxone (Experimental)
  Interventions: Drug: naloxone
- normal saline (Placebo Comparator)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: naloxone — 10 mg naloxone in 25 ml total volume
  Other Names: endorphin receptor antagonist
  Arms: naloxone
Drug: normal saline — 25 ml
  Other Names: salt water
  Arms: normal saline

SUMMARY:
Endorphins are released in response to breathing difficulty and can modify the perception of breathlessness. In this randomized placebo-controlled trial, resistive breathing loads are used to provoke breathlessness in patients with chronic obstructive pulmonary disease. The hypothesis of the study is that intravenous (IV) administration of naloxone, a medication which blocks endorphin activity, will increase the perception of breathlessness experienced by patients while breathing through a resistance device, compared with IV administration of normal saline.

DETAILED DESCRIPTION:
Study Design:

The study is a randomized, double-blind, placebo-controlled investigation comparing the intravenous administration of:

* normal saline, considered a placebo, is expected to have no effect on patient ratings of dyspnea.
* naloxone, an opioid receptor antagonist with penetration into the central nervous system and blocks the effect of beta-endorphins, is expected to increase ratings of dyspnea in patients with COPD.

Dyspnea will be induced by resistive load breathing for a minimum of 10 minutes.

Subjects:

Twenty subjects with COPD will be recruited from the outpatient clinic at the Dartmouth-Hitchcock Medical Center.

Procedures:

There are three visits each 2 - 3 days apart.

Visit 1

The purposes of Visit 1 are:

* to ensure that patients meet inclusion and exclusion criteria
* to collect baseline data
* to familiarize each patient with the study protocol
* to practice breathing through the resistive load system

Visit 2 (2 - 3 days after Visit 1)

Patients will perform pulmonary function tests and then inhale 2 puffs (180 mcg) of albuterol metered-dose inhaler (MDI) in order to provide standardized bronchodilatation prior to resistance breathing. Thirty minutes later, pulmonary function tests will be repeated to measure the response.

Next, patients will be randomized to one of two blinded study medications.

1. normal saline (25 ml volume) intravenous infusion given 5 minutes before resistive breathing
2. naloxone (10mg in 25 ml total volume) intravenous push given 5 minutes prior to resistive breathing

An 18-20 gauge catheter will be inserted into an arm vein to be used for drawing blood and for administration of either normal saline or naloxone. In a seated position, the patient will breathe quietly through the mouth piece without any resistance. After 5 minutes, 10 ml of venous blood will be removed for measurement of baseline plasma beta-endorphin immunoreactivity. Then, the physician will give the normal saline or naloxone solution intravenously through tubing connected to the catheter. Five minutes after the infusion has been given, the resistance load (obtained at Visit 1) will be added to the inspiratory side of a two-way valve. The patient will be instructed to continue breathing through the resistance "for as long as possible." At one minute intervals, the patient will be asked to place a mark on a vertical visual analog scale (VAS) in order to rate separately the intensity and the unpleasantness of dyspnea. When the patient is no longer able to breathe through the resistance system, the patient will be asked to make final ratings of the intensity and the unpleasantness of dyspnea. Thereafter, resistance breathing will be stopped, and the mouthpiece will be removed from the patient. Next, 10ml of venous blood will be removed for measurement of the plasma beta-endorphin immunoreactivity. A third 10 ml aliquot of venous blood will be taken at 30 minutes after completion of the resistive breathing session.

During the 5 minutes of breathing normally at rest and during the resistance breathing, the following non-invasive measurements will be made: inspiratory mouth pressure (Pm); expired gas will be analyzed breath-by-breath for minute ventilation (VE), oxygen consumption (VO2), and carbon dioxide production (VCO2) using a metabolic measurement system (MedGraphics); oxygen saturation will be recorded using a pulse oximeter; and end-tidal partial pressure of CO2.

Visit 3

At Visit 3, the same procedures will be used as described for Visit 2, except that the patient will be randomized to the alternative blinded study medication that he/she did not receive at Visit 2.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient 50 years of age or older;
* A diagnosis of COPD defined by American Thoracic Society-European Respiratory Society criteria
* Current or former smoker with a smoking history of greater than or equal to 10 pack-years;
* A post-bronchodilator forced expiratory volume in one second (FEV1) greater than or equal to 30% predicted and less than or equal to 80% predicted; AND
* A post-bronchodilator FEV1/forced vital capacity ratio less than 70%; and clinically stable COPD.

Exclusion Criteria:

* Any patient who has a concomitant disease that might interfere with study procedures or evaluation;
* Inability to perform resistive breathing maneuvers; OR
* Any current use of a narcotic medication.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald A Mahler, M.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Result] Gifford AH, Mahler DA, Waterman LA, Ward J, Kraemer WJ, Kupchak BR, Baird JC. Neuromodulatory effect of endogenous opioids on the intensity and unpleasantness of breathlessness during resistive load breathing in COPD. COPD. 2011 Jun;8(3):160-6. doi: 10.3109/15412555.2011.560132. Epub 2011 Apr 22. PMID 21513438

RESULTS

PARTICIPANT FLOW:
Recruitment Details: March 2009 - June 2010; medical center
Pre-assignment Details: 17 subjects recruited; 3 subjects excluded (2 did not meet inclusion criteria; 1 refused participation after signing consent).
Groups:
- Normal Saline First, Then Naloxone: Intravenous saline (25 ml) in first intervention period and intravenous Naloxone (10mg/25 ml) in second intervention period.
- Naloxone First, Then Normal Saline: Intravenous Naloxone (10mg/25 ml)in first intervention period and intravenous saline (25 ml) in second intervention period.
Period: First Intervention
Arm/Group | Normal Saline First, Then Naloxone | Naloxone First, Then Normal Saline
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Normal Saline First, Then Naloxone | Naloxone First, Then Normal Saline
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive saline first and Naxolone first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 64 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Intensity of Breathlessness
Description: The average of all ratings for the intensity of breathlessness at equivalent times for each subject during Resistive Load Breathing (RLB). For example, if 1 subject provided 6 ratings during 6 minutes of RLB with naloxone and 10 ratings during 10 minutes of RLB with normal saline, then ratings for intensity through 6 minutes were used for analysis for that patient. This approach was used for all subjects to yield a total of 154 ratings for naloxone and for normal saline.
  Subject rating of intensity of breathlessness was obtained at 1 minute intervals during RLB on a 100 mm Visual Analog Scale anchored at the bottom by "No Intensity" and at the top by "Greatest Intensity".
Time Frame: At 1 minute intervals during Resistive Load Breathing at Period 1 (Day 3 or 4) and Period 2 (Day 5, 6 or 7)
Population: Total number of subjects completing both periods of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Normal Saline: Intravenous saline (25 ml)
- Naloxone: Intravenous Naloxone (10mg/25ml)
Arm/Group | Normal Saline | Naloxone
Number analyzed (Participants) | 14 | 14
units on a scale | 77 (21) | 83 (18)
Statistical Analysis 1: Comparison: Normal Saline vs Naloxone; Test type: Superiority or Other; p = .0004, t-test, 2 sided; Mean Difference (Net) = 5, 95% CI 2-sided [2.69 to 9.38]

2. Primary Outcome: Unpleasantness of Breathlessness
Description: The average of all ratings for the unpleasantness of breathlessness at equivalent times for each subject during Resistive Load Breathing (RLB). For example, if 1 subject provided 6 ratings during 6 minutes of RLB with naloxone and 10 ratings during 10 minutes of RLB with normal saline, then ratings for intensity through 6 minutes were used for analysis for that patient. This approach was used for all subjects to yield a total of 154 ratings for naloxone and for normal saline.
  Subject rating of intensity of unpleasantness was obtained during RLB on a 100 mm Visual Analog Scale anchored at the bottom by "No Unpleasantness" and at the top by "Greatest Unpleasantness".
Time Frame: At 1 minute intervals during Resistive Load Breathing at Period 1 (Day 3 or 4) and Period 2 (Day 5, 6 or 7)
Population: Total number of subjects completing both periods of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Naloxone: Intravension Naloxone (10mg/25ml)
Arm/Group | Normal Saline | Naloxone
Number analyzed (Participants) | 14 | 14
units on a scale | 77 (19) | 81 (20)
Statistical Analysis 1: Comparison: Normal Saline vs Naloxone; Test type: Superiority or Other; p = .024, t-test, 2 sided; Mean Difference (Net) = 4, 95% CI 2-sided [0.49 to 6.85]

3. Secondary Outcome: Endurance Time
Description: Length of time that subjects were able to continue Resistive Load Breathing
Time Frame: Period 1 (Day 3 or 4) and Period 2 (Day 5, 6 or 7)
Population: Total number of subjects completing both periods of the study.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Normal Saline: Intravenous saline (25 ml) given prior to start of Resistive Load Breathing
- Naloxone: Intravenous Naloxone (10mg/25ml)given prior to start of Resistive Load Breathing
Arm/Group | Normal Saline | Naloxone
Number analyzed (Participants) | 14 | 14
minutes | 13.9 (4.7) | 12.5 (5.4)
Statistical Analysis 1: Comparison: Normal Saline vs Naloxone; Test type: Superiority or Other; p = 0.45, t-test, 2 sided

4. Secondary Outcome: Change in Level of B-endorphin Immunoreactivity During Naloxone Intervention
Description: Change in serum levels of beta-endorphin immunoreactivity measured in pmol/L in subjects receiving Naloxone
Time Frame: Baseline and at the end of Resistance Load Breathing during either Period 1 (Day 3 or 4) or Period 2 (Day 5, 6 or 7) depending on randomization
Population: Total number of subjects completing period with Naloxone intervention.
Measure: Mean (Standard Deviation); unit: pmol/L
Groups:
- Baseline: Pre-infusion of Naloxone (10 mg/25 ml)
- End of Resistance Load Breathing: End of Resistance Load Breathing post-infusion of Naloxone (10 mg/25 ml)
Arm/Group | Baseline | End of Resistance Load Breathing
Number analyzed (Participants) | 14 | 14
pmol/L | 6.0 (1.5) | 18.5 (3.4)
Statistical Analysis 1: Comparison: Baseline vs End of Resistance Load Breathing; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

5. Secondary Outcome: Change in Level of B-endorphin Immunoreactivity During Saline Intervention
Description: Change in serum levels of beta-endorphin immunoreactivity measured in pmol/L in subjects receiving Saline
Time Frame: as for outcome 4
Population: Total number of subjects completing period with saline intervention.
Measure: Mean (Standard Deviation); unit: pmol/L
Groups:
- Baseline: Pre-infusion of Normal Saline (25 ml)
- End of Resistance Load Breathing: End of Resistance Load Breathing post-infusion of Normal Saline (25 ml)
Arm/Group | Baseline | End of Resistance Load Breathing
Number analyzed (Participants) | 14 | 14
pmol/L | 6.7 (1.4) | 13.4 (2.5)
Statistical Analysis 1: Comparison: Baseline vs End of Resistance Load Breathing; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- Normal Saline: 25 ml Intravenous
- Naloxone: 10mg/25ml Intravenous
Arm/Group | Normal Saline | Naloxone
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No